CLINICAL TRIAL: NCT04645979
Title: The Perception of Celestamine Treatment in Mexico: a Retrospective Assessment of Consumer Perception of Prior Celestamine Use
Brief Title: A Study to Learn What Participants Think of Treatment With Betamethasone Plus Loratadine to Treat Their Acute Allergic Rhinitis, Also Known as Hay Fever in Mexico
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21614
Record Dates: First submitted 2020-11-23; First posted 2020-11-27 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants who used betamethasone plus loratadine to treat allergic rhinitis within the previous two months.
  Interventions: Other: Online survey

INTERVENTIONS:
Other: Online survey — Participants will be invited to complete an online questionnaire about their experience of product use.

SUMMARY:
Acute allergic rhinitis is a common allergic reaction to things like pollen or dust. It causes inflammation inside the nose, resulting in symptoms similar to the common cold. Allergic rhinitis is also known as hay fever.

In this study, the researchers want to learn what participants think of betamethasone plus loratadine as a treatment for their acute allergic rhinitis. These participants will have used betamethasone plus loratadine as a treatment for their acute allergic rhinitis within the past two months. During the study, participants will complete an online questionnaire about their experience with betamethasone plus loratadine.

ELIGIBILITY:
Inclusion Criteria:

* Participants who used betamethasone plus loratadine within the previous 2 months for the treatment of acute episodes of allergic rhinitis
* Participants allowing to use the data for research and marketing purposes as well as talking to authorities
* Participants allowing us to use the pseudo-randomized individual data for further data analysis
* Able to read and understand the language of the online questionnaire

Exclusion Criteria:

- None

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population are participants who used betamethasone plus loratadine within the previous 2 months for the treatment of acute episodes of allergic rhinitis.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Experience with betamethasone plus loratadine via an online questionnaire | 2 months
  Participants' experiences with betamethasone plus loratadine used under real life conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Mexico

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/